CLINICAL TRIAL: NCT03746171
Title: Blue Light Imaging (BLI) for Optical Diagnosis of Colorectal Polyps: the BLI Resect and Discard (BIRD) Study.
Brief Title: Blue Light Imaging (BLI) for Optical Diagnosis of Colorectal Polyps
Acronym: BIRD
Status: Completed | Type: Observational
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Franco Radaelli, Head of Gastrointestinal Endoscopy Unit, Valduce Hospital
Other Study IDs: 229
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Colonic Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with rectosigmoid colonic polyps: Consecutive adult (18-80 yrs) outpatients undergoing colonoscopy in the frame of the FOBT based screening program, in which at least one diminutive (<5 mm) rectosigmoid polyp is detected.
  Interventions: Diagnostic Test: Colonic polyp characterization by BLI

INTERVENTIONS:
Diagnostic Test: Colonic polyp characterization by BLI — All rectosigmoid <5 mm polyps, regardless of the presence of larger polyps, will be characterized by BLI-assisted optical diagnosis by using BASIC criteria (neoplastic vs. non neoplastic) and will be included in polyp-level assessment.
  The polyp characterization will be always performed and recorded without zoom magnification. In patients in which colonoscopy will be performed with endoscopes equipped with zoom magnification, the zoom will be eventually systematically applied and the characterization with zoom will be also recorded. The post-polypectomy surveillance intervals based on BLI will be calculated by using histology estimation performed without zoom for all patients. Only polyps characterized with high confidence will be included in the analysis; the high-confidence characterization rate will be calculated.

SUMMARY:
Several imaging technologies have been developed in order to enable the endoscopists to differentiate neoplastic from non-neoplastic lesions. The real-time prediction of polyps histology is clinically relevant as diminutive polyps represent the majority of polyps detected during colonoscopy and have a very low risk of harboring advanced histology or invasive carcinoma. Thus, an optical diagnosis would allow diminutive polyps to be resected and discarded without pathological assessment or left in place without resection, with an enormous cost-saving potential. Recently, the American Society of Gastrointestinal Endoscopy (ASGE) has set the Preservation and Incorporation of Valuable endoscopic Innovation (PIVI) which defined accuracy threshold to be met, in order to consider a new technology ready to be incorporate into clinical practice. Blue Light Imaging (BLI) is a new chromoendoscopy technology integrated in the latest generation ELUXEOTM 7000 endoscopy platform (Fujifilm Co, Tokyo, Japan), based on the direct (i.e. not filtered) emission of blue light with short wavelength (410nm), that enhances visibility of both microvascular and superficial mucosal pattern. In a recent randomized trial BLI was superior to high-definition white light (HDWL) in the real time characterization of subcentimetric and diminutive colonic polyps. Nevertheless, in this study the paucity of diminutive rectosigmoid polyps analyzed does not allow to draw definite conclusions as the meeting of PIVI thresholds are concerned. Similarly, the low numbers of patients evaluated limited the per-patient analysis. Therefore further studies adequately powered to this clinically end-point were advocated. Additionally, when the study was performed a BLI dedicated classification for optical diagnosis of colonic polyps was not available, whereas recently a specific classification (the BLI Adenoma Serrated International Classification-BASIC) has been developed and a specific training set has been settled.

In the present study the investigators prospectively evaluate whether the use of BLI-assisted optical characterization of diminutive polyps using BASIC classification by specifically trained endoscopists may met PIVI thresholds and particularly if it allow the endoscopists to achieve > 90% correct assignment of post-polypectomy surveillance intervals when combined with the histopathology assessment of polyps >5 mm in size.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult (18-80 yrs) outpatients undergoing colonoscopy in the frame of the FOBT based screening program or for CRC primary prevention, in which at least one diminutive (<5 mm) rectosigmoid polyp is detected.

Exclusion Criteria:

* patients with CRC history or hereditary polyposis syndromes or hereditary non-polyposis colorectal cancer
* patients with inadequate bowel preparation
* patients in which caecal intubation was not achieved or scheduled for partial examinations
* polyps could not be resected due to ongoing anticoagulation preventing resection and pathologic assessment

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive adult (18-80 yrs) outpatients undergoing colonoscopy in the frame of the FOBT based screening program or for CRC primary prevention, in which at least one diminutive (<5 mm) rectosigmoid polyp is detected.
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of post-polypectomy surveillance interval | 9 months
  Surveillance interval will be advised for each patient, basing on high-confidence predictions of <5mm polyp histology. Such information will be merged with the histopathology assessment of both polyps >5 mm in size and <5 mm lesions diagnosed with a low confidence. Patients with either only <5 mm lesions diagnosed with a low confidence or only >6 mm lesions will not be included. Endoscopy-directed surveillance strategy will be subsequently matched with histology-directed one for each patient and accordance rate will be calculated.
  The post-polypectomy surveillance interval will be calculated in the frame of USMSTF guidelines.

SECONDARY OUTCOMES:
Accuracy parameters of BLI polyp characterization | 9 months
  Operative characteristics (sensitivity, specificity, positive and negative predictive value and accuracy) in distinguishing adenomatous from non-adenomatous polyps, evaluated with high confidence, will be calculated for each diminutive rectosigmoid polyp, having histopathology report as reference standard.
Cost analysis | 9 months
  The cost (related to the polypectomy devices used and the histopathology assessment) will be calculated according to a BLI-directed policy and to a histology-directed policy per each patient included in the study. The cost saving will be eventually calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Radaelli, MD, Principal Investigator — Valduce Hospital
Locations (1):
- Ospedale Valduce, Como, Italy

REFERENCES:
- [Derived] Rondonotti E, Hassan C, Andrealli A, Paggi S, Amato A, Scaramella L, Repici A, Radaelli F. Clinical Validation of BASIC Classification for the Resect and Discard Strategy for Diminutive Colorectal Polyps. Clin Gastroenterol Hepatol. 2020 Sep;18(10):2357-2365.e4. doi: 10.1016/j.cgh.2019.12.028. Epub 2020 Jan 7. PMID 31923641